CLINICAL TRIAL: NCT03705481
Title: CorPath GRX With ReMOTE Proof of Principle (POP): First in Human in India
Brief Title: GRX With ReMOTE: First in Human in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 104-07972
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, single center, non-randomized feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Remote treatment of PCI. (Other): 5 sequential subjects presenting for remote PCI who have signed informed consent.
  Interventions: Device: Remote treatment of PCI.

INTERVENTIONS:
Device: Remote treatment of PCI. — To evaluate the safety and performance of CorPath GRX POP System, in the ReMOTE (location outside hospital) delivery and manipulation of coronary guidewires and stent/balloon catheters, and manipulation of guide catheters during PCI procedures.
  Other Names: CorPath GRX and Proof of Principle System

SUMMARY:
To evaluate the safety and performance of CorPath GRX POP System, in the ReMOTE (location outside hospital) delivery and manipulation of coronary guidewires and stent/balloon catheters, and manipulation of guide catheters during PCI procedures.

DETAILED DESCRIPTION:
Prospective, single-arm, single center, non-randomized feasibility study of the CorPath GRX POP System to examine its performance during remote angioplasty (ballooning) and stenting and patient outcomes through 48 hours post-PCI procedure hospital discharge, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients with coronary artery disease with clinical indication for PCI;
3. Patient deemed appropriate for robotic-assisted PCI; and
4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Angiographic Inclusion:

1. Study lesion is a single de novo native coronary artery lesion (i.e. a coronary lesion not previously treated).
2. The lesion reference vessel diameter is between 2.50 mm and 4.0 mm by visual estimate.
3. Study lesion length less or equal to 20 mm by visual estimate.
4. The study lesion length can be treated with one stent. The stent should be able to cover the whole length of the lesion with at least 2 mm of normal segments on proximal and distal edges of the lesion.
5. Study lesion diameter showing significant stenosis of at least 50% by visual estimate.

Exclusion Criteria:

1. Failure/inability/unwillingness to provide informed consent; or
2. The investigator determines that the patient or the coronary anatomy is not suitable for robotic-assisted PCI.

Angiographic Exclusion:

1. Target lesion that cannot be fully covered by a single stent.
2. Subject requires treatment of multiple lesions
3. Any previous stent placement within 5 mm (proximal or distal) of the target lesion
4. The study lesion requires planned treatment with DCA, laser, rotational atherectomy, or any device except for balloon dilatation prior to stent placement
5. The study vessel has evidence of intraluminal thrombus or moderate to severe tortuosity (> 90°) proximal to the target lesion
6. The study lesion has any of the following characteristics:

   1. Total occlusion
   2. Within 2mm of a side branch > 2.0 mm vessel diameter
   3. Not ostial in location
   4. Is located at ≥ 45° bend in the vessel
   5. Is severely tortuous
   6. Is severely calcified
   7. Severe calcification at the part of the vessel proximal to target lesion
   8. Target lesion that is located in a native vessel distal to an anastomosis with a saphenous vein graft or a left/right internal mammary artery (LIMA/RIMA) bypass and is approached through the by-pass graft
7. Unprotected left main coronary artery disease (an obstruction greater than 50% diameter stenosis in the left main coronary artery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tejas Patel, MD, Principal Investigator — Apex Heart Institute
Locations (1):
- Apex Heart Institute, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Madder RD, VanOosterhout SM, Jacoby ME, Collins JS, Borgman AS, Mulder AN, Elmore MA, Campbell JL, McNamara RF, Wohns DH. Percutaneous coronary intervention using a combination of robotics and telecommunications by an operator in a separate physical location from the patient: an early exploration into the feasibility of telestenting (the REMOTE-PCI study). EuroIntervention. 2017 Jan 20;12(13):1569-1576. doi: 10.4244/EIJ-D-16-00363. PMID 28105993
- [Result] Pugin F, Bucher P, Morel P. History of robotic surgery: from AESOP(R) and ZEUS(R) to da Vinci(R). J Visc Surg. 2011 Oct;148(5 Suppl):e3-8. doi: 10.1016/j.jviscsurg.2011.04.007. Epub 2011 Oct 4. No abstract available. PMID 21974854
- See also: Surgeons perform transatlantic operation using fibreoptics — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1121281/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Remote Treatment of PCI.
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 5 participants in the study.
Groups:
- Age at Time of Consent: Age at the time of consent for the subjects that had a CorPath robotic PCI procedure performed remotely.
Arm/Group | Age at Time of Consent
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] — Participants whose age is > 18 years.
  years | 54 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Device Technical Success
Description: Defined as completing the robotic PCI entirely with the CorPath GRX POP System.
Time Frame: Measured from guide catheter in time through procedure end time (or guide catheter out time).
Population: Number of participants that had a remote robotic assisted PCI without unplanned conversion to manual technique.
Measure: Count of Participants; unit: Participants
Groups:
- Device Technical Success: Number of participants that had a successful completion of the ReMOTE robotic-assisted PCI absent unplanned conversion to manual.
Arm/Group | Device Technical Success
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: In-hospital MACE
Description: Recording any MACE event that occurred from the time the sheath was inserted through 48 hours post procedure or hospital discharge, whichever of the two occurred first.
Time Frame: Measured from Sheath in time to discharge or 48 hours, whichever occurs first.
Population: Number of participants with an In-hospital MACE occurrence.
Measure: Count of Participants; unit: Participants
Groups:
- In-hospital MACE: MACE that occurs within 48 hours of the procedure or prior to hospital discharge, whichever occurs first, in a subject treated with CorPath GRX.
Arm/Group | In-hospital MACE
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Clinical Procedural Success
Description: Number of patients with a residual stenosis (visual estimate, less than 30%) post PCI in the lesion(s) treated with the CorPath GRX POP System.
Time Frame: Measured from guide catheter in time through procedure end time (or guide catheter out time).
Population: Number of participants with a residual stenosis less than 30% (visual estimate).
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Procedural Success: Defined as less than 30% residual stenosis (visual estimate) post PCI in the lesion(s) treated with the CorPath GRX POP System
Arm/Group | Clinical Procedural Success
Number analyzed (Participants) | 5
Participants | 5

4. Secondary Outcome: All Serious Adverse Events
Description: Recording any SAE that occurred measured from the sheath insertion time through 48 hours post procedure or hospital discharge, whichever occurred first.
Time Frame: Measured from Sheath in time to discharge or 48 hours, whichever occurs first.
Population: Number of participants with a Serious Adverse Events (SAEs) from the start of the Re- MOTE CorPath procedure until the end of the study
Measure: Count of Participants; unit: Participants
Groups:
- All Serious Adverse Events: ll Serious Adverse Events (SAEs) from the start of the Re- MOTE CorPath procedure until the end of the study.
Arm/Group | All Serious Adverse Events
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: MACE that occurs within 48 hours of the procedure or prior to hospital discharge.
Description: Major Adverse Cardiac Event (MACE): MACE is defined as cardiac death, Q-wave or non-Q-wave myocardial infarction (MI), or clinically driven target vessel revascularization (TVR) by per-cutaneous or surgical methods.
  Serious Adverse Events - all serious adverse events that were collected during the study, whether or not they were anticipated or considered to be attributed or associated with the intervention.
Arm/Group | Remote Treatment of PCI.
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03705481/Prot_SAP_001.pdf